CLINICAL TRIAL: NCT06326437
Title: The Effects of Dyadic Intervention for Young and Middle-aged Couples Facing Colorectal Cancer: A Randomised Controlled Trial
Brief Title: Dyadic Intervention for Psychological Distress of Patients With Colorectal Cancer and Their Spouses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Qian Sun, PhD student, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1223
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 6-week dyadic intervention (Experimental): A 6-week psychosocial dyadic programme comprises 6 weekly 60-90min internet-based sessions.
  Interventions: Other: 6-week dyadic intervention
- Usual care (No Intervention): The control group to receive the usual care provided by the clinical team in the hospital.

INTERVENTIONS:
Other: 6-week dyadic intervention — Comprising 6 weekly 60-90min internet-based sessions.
  Arms: 6-week dyadic intervention

SUMMARY:
The overall aim of the study is to evaluate the effects of a dyadic intervention on mutuality, psychological strengths (i.e., illness cognition and dyadic coping), illness-related communication, psychological distress, and QoL outcomes of patients with colorectal cancer and spouses. The colorectal cancer couples were randomly allocated to the intervention group to receive a 6-week dyadic intervention, or to the control group to receive the usual care provided by the clinical team in the hospital.

ELIGIBILITY:
Inclusion Criteria:

patients and spouses aged 20 years or older patients diagnosed with colorectal cancer within the past year Patients scored ≥ 22 points on the Kessler Psychological Distress Scale assessment patients and spouses able to read simplified Chinese

Exclusion Criteria:

psychiatric problems requiring active treatment other terminal illnesses, such as advanced cancer currently undergoing psychotherapy or participating in similar trials

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
the Kessler psychological distress scale-10 | Changes from baseline (T0) to immediately (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after the intervention
  The scale employs a Likert 5-point rating system, ranging from "almost never" to "all the time" with values assigned from 1 to 5 respectively, yielding a total score between 10 and 50. Higher scores indicate greater levels of psychological distress, with a cutoff set at ≥22 points.

SECONDARY OUTCOMES:
The Illness Cognition Questionnaire | Changes from baseline (T0) to immediately (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after the intervention
  The Chinese version of the Illness Cognition Questionnaire comprises three dimensions: helplessness, acceptance, and perceived benefits, each featuring six items, totaling 18 items. It employs a Likert 4-point rating scale, ranging from "completely disagree" to "completely agree." Each dimension is scored independently, with scores ranging from 6 to 24. Higher scores indicate a heightened perception within the respective dimension, and scores from different dimensions are not aggregated.
Dyadic Coping Inventory | Changes from baseline (T0) to immediately (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after the intervention
  The scale is designed to evaluate partners' joint coping behaviors in response to shared sources of stress. It utilizes a Likert 5-point rating system, where 1 represents "rarely" and 5 represents "very frequently." Notably, items 7, 10, 11, 15, 22, 25, 26, and 27 are reverse-scored. Additionally, items 36 and 37 assess self-rated satisfaction with binary strategy use and are excluded from the total score calculation. The overall Cronbach's α coefficient for the scale is 0.92, with individual dimension coefficients ranging from 0.67 to 0.91.
European Organization for Research and Treatment of Cancer, Quality of Life Questionnaire-Core 30 | Changes from baseline (T0) to immediately (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after the intervention
  The scale, developed by the European Organization for Research and Treatment of Cancer, consists of 30 items. It evaluates five functional domains (physical, emotional, cognitive, social, and role functioning), nine symptom domains (nausea and vomiting, diarrhea, constipation, fatigue, pain, insomnia, appetite loss, dyspnea, and financial difficulties), and one overall health status domain. Scores range from 0 to 100, with higher scores indicating better quality of life. The Cronbach's α coefficient for the overall quality of life scale is 0.809.
Locke-Wallace Marital Adjustment Scale | Changes from baseline (T0) to immediately (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after the intervention
  Locke-Wallace Marital Adjustment Scale was used to measure marriage quality. Total score was 0-158 points, although higher scores suggest better marriage quality.
Mutual communication | Changes from baseline (T0) to immediately (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after the intervention
  Cancer- Related Communication Problems within Couple Scale (CRCP) is a 15- item measure assessing cancer- related communication problems within a cancer couple (e.g. 'My spouse does not ask how cancer affected my life' for patients, and 'My spouse does not ask about how him/her having cancer affects my life' for SCs; Kornblith et al., 2006). Higher scores demonstrate more communication problems within a cancer couple. Coefficient alpha in Chinese cancer patients and their SCs were .805 and .737, respectively (Li et al., 2015).
Caregiving burden | Changes from baseline (T0) to immediately (T1), 1 month (T2), 3 months (T3), and 6 months (T4) after the intervention
  The Zarit Burden Inventory (Zarit Burden Inventory, ZBI) (Appendix 8) was used to assess the care burden of spouses of colorectal cancer patients. This scale was introduced by Wang Lie et al. [227] in 2006. It consists of 22 items and assesses the social life, economic status, mental status and health status of the primary caregivers in four aspects. The total score ranges from 0 to 88 points. The higher the score, the heavier the care burden. The Cronbach's α coefficient of this scale is 0.87

CONTACTS AND LOCATIONS:
Overall Officials: Qian Sun, PhD student, Principal Investigator — Sun Yat-sen Univesity
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No